CLINICAL TRIAL: NCT00949442
Title: Superiority of Insulin Glargine Lantus vs. NPH: Treat to Normoglycemia Concept.Effect of Insulin Glargine in Comparison to Insulin NPH in Insulin-nave People With Type 2 Diabetes Mellitus Treated With at Least One OAD and Not Adequately Controlled
Brief Title: Lantus Versus NPH: Comparison in Insulin Naive People Not Adequately Controlled With at Least One Oral Anti Diabetics (OAD) Treatment
Acronym: LANCELOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_C_02762; EUDRACT #: 2007-006640-22
Record Dates: First submitted 2009-07-27; First posted 2009-07-30 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; glimepiride; Insulin, Isophane

ARMS (2):
- 1 (Experimental): Before randomization (common with arm 2):
  2 weeks of Screening phase: Oral Anti Diabetics (OAD) 2 weeks of Run-In phase: switch of OAD (Sulfonylurea (except Glimepiride), glinides or alpha-glucosidase inhibitor) to Glimepiride
  After randomization:
  36 weeks of study treatment phase: Insulin Glargine + OAD(s) at stable dose
  Interventions: Drug: Insulin Glargine (HOE901) [Lantus]; Drug: Glimepiride
- 2 (Active Comparator): Before randomization (common with arm 1):
  2 weeks of Screening phase: Oral Anti Diabetics (OAD) 2 weeks of Run-In phase: switch of OAD (Sulfonylurea (except Glimepiride), glinides or alpha-glucosidase inhibitor) to Glimepiride
  After randomization:
  36 weeks of study treatment phase: NPH + OAD(s) at stable dose
  Interventions: Drug: Glimepiride; Drug: human insulin [NPH]

INTERVENTIONS:
Drug: Insulin Glargine (HOE901) [Lantus] — 100 Units/ml solution for injection in a pre-filled pen SoloStar® (3 ml)
  Arms: 1
Drug: Glimepiride — tablets of 1 and 2 mg
Drug: human insulin [NPH] — 100 IU/ml suspension for injection in a prefilled pen OptiSet® (3 ml)
  Arms: 2

SUMMARY:
Primary Objective:

To demonstrate the superiority of insulin glargine over insulin NPH (Neutral Protamin Hagedornon) the change in HbA1c from baseline to the end of the treatment period.

Secondary Objective:

To compare between treatment groups:

* Plasma glucose (fasting, nocturnal) over time,
* Changes from baseline in HbA1c over time,
* Percentage of patients who reach the target of HbA1c <7 and <6.5,
* Use of prandial insulin as rescue medication at month 6,
* Incidence and rate of hypoglycemia (symptomatic diurnal and nocturnal, asymptomatic and severe),
* Daily dose of insulin,
* Change in body weight from baseline,
* Evolution of 8-point plasma-glucose (PG) profiles,
* Overall safety,
* Patient reported outcomes (treatment satisfaction).

ELIGIBILITY:
Inclusion Criteria

* Insulin-naïve type 2 diabetes mellitus
* Type 2 diabetes mellitus diagnosed for at least 1 year
* Treated with at least one OAD (Metformin [daily dose of at least 1000mg], Sulfonylurea, glinides or alpha-glucosidase inhibitor) at stable dose for at least 3 months.
* HbA1c > or = 7.0% and < or = 10.5%
* BMI < 40 kg/m²
* Ability and willingness to perform plasma glucose monitoring using the sponsor-provided glucose meter and patient diary at home
* Informed consent obtained in writing at enrolment into the study
* Willingness and ability to comply with the study protocol

Exclusion criteria:

* Treatment with GLP-1 agonists or with DPP-IV inhibitors in the 3 months prior to study entry
* Treatment with TZD as monotherapy
* Diabetes mellitus other than Type 2 (e.g. secondary to pancreatic disorders, drugs or chemical agents intake...)
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study (an optic fundus examination should have been performed within the 2 years prior to study entry)
* Impaired renal function: serum creatinine > or =1.5 mg/dL (> or = 133µmol/L) or > or = 1.4 mg/dL (> or = 124 µmol/L) in men and women, respectively
* History of sensitivity to the study drugs or to drugs with a similar chemical structure
* Impaired hepatic function (ALT and/or AST > 3 x upper limit of normal range)
* Pregnant or lactating women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method),
* Treatment with systemic corticosteroids within the 3 months prior to study entry or likelihood of requiring treatments during the study which are not permitted.
* Treatment with an investigational product in the 30 days prior to visit 1
* Alcohol or drug abuse in the last year
* Presence of any condition (medical, psychological, social or geographical), current or anticipated that the Investigator feels would compromise the patient's safety or limit the patient successful participation in the study (including night shift worker)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | Recorded at baseline (week 0), week 12, week 24 and week 36

SECONDARY OUTCOMES:
Self-monitored fasting plasma glucose (FPG) | Before baseline (week 0), weeks 12, 24 and 36
8-points profiles | The week before baseline, at 12, 24 and 36 weeks
Episodes of hypoglycemia | From the week -2 to the week 36
Daily doses of insulin | At week 1, week 2, week 3, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 20, week 24, week 28, week 32, week 36
Need of additional prandial insulin | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Pilorget, MD, Study Director — Sanofi
Locations (87):
- Brazil (7):
  - Investigational Site Number 076-001, Fortaleza
  - Investigational Site Number 076-006, Fortaleza
  - Investigational Site Number 076-005, Porto Alegre
  - Investigational Site Number 076-007, Rio de Janeiro
  - Investigational Site Number 076-004, São Paulo
  - Investigational Site Number 076-003, São Paulo
  - Investigational Site Number 076-002, São Paulo
- Czechia (11):
  - Investigational Site Number 203003, Beroun
  - Investigational Site Number 203001, Chrudim III
  - Investigational Site Number 203008, České Budějovice
  - Investigational Site Number 203011, České Budějovice
  - Investigational Site Number 203006, Hodonín
  - Investigational Site Number 203002, Hranice I - Mesto
  - Investigational Site Number 203010, Liberec
  - Investigational Site Number 203009, Moravský Písek
  - Investigational Site Number 203004, Prague
  - Investigational Site Number 203005, Prague
  - Investigational Site Number 203007, Prague
- Investigational Site Number 818001, Menoufiya, Egypt
- France (6):
  - Investigational Site Number 250-002, Aix-en-Provence
  - Investigational Site Number 250-001, Antibes
  - Investigational Site Number 250-005, Bordeaux
  - Investigational Site Number 250-004, Jarny
  - Investigational Site Number 250-003, Narbonne
  - Investigational Site Number 250-006, Strasbourg
- Investigational Site Number 380001, Perugia, Italy
- Investigational Site Number 414001, Kuwait City, Kuwait
- Mexico (6):
  - Investigational Site Number 484003, Guadalajara
  - Investigational Site Number 484005, Guadalajara
  - Investigational Site Number 484001, Monterrey
  - Investigational Site Number 484008, Pachuca
  - Investigational Site Number 484009, Pachuca
  - Investigational Site Number 484002, Puebla City
- Netherlands (6):
  - Investigational Site Number 528006, Almelo
  - Investigational Site Number 528005, Apeldoorn
  - Investigational Site Number 528001, Beek
  - Investigational Site Number 528002, Hoogeveen
  - Investigational Site Number 528004, Hoogezand
  - Investigational Site Number 528003, Rotterdam
- Poland (4):
  - Investigational Site Number 616004, Gdansk
  - Investigational Site Number 616003, Krakow
  - Investigational Site Number 616002, Lublin
  - Investigational Site Number 616001, Zabrze
- Romania (11):
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642009, Cluj-Napoca
  - Investigational Site Number 642003, Craiova
  - Investigational Site Number 642005, Iași
  - Investigational Site Number 642010, Oradea
  - Investigational Site Number 642011, Oradea
  - Investigational Site Number 642007, Ploieşti
  - Investigational Site Number 642004, Reşiţa
  - Investigational Site Number 642008, Târgu Mureş
  - Investigational Site Number 642012, Timișoara
- Russia (7):
  - Investigational Site Number 643-001, Moscow
  - Investigational Site Number 643-002, Saint Petersburg
  - Investigational Site Number 643-003, Saint Petersburg
  - Investigational Site Number 643-006, Samara
  - Investigational Site Number 643-005, Saratov
  - Investigational Site Number 643-004, St-Ptetersburg
  - Investigational Site Number 643-007, Tyumen
- Slovakia (8):
  - Investigational Site Number 703005, Banská Bystrica
  - Investigational Site Number 703003, Bratislava
  - Investigational Site Number 703007, Bratislava
  - Investigational Site Number 703004, Košice
  - Investigational Site Number 703006, Košice
  - Investigational Site Number 703002, Košice
  - Investigational Site Number 703008, Levice
  - Investigational Site Number 703001, Martin
- South Korea (6):
  - Investigational Site Number 410005, Daegu
  - Investigational Site Number 410002, Gyeonggi-do
  - Investigational Site Number 410006, Incheon
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410004, Seoul
- Sweden (4):
  - Investigational Site Number 752004, Lund
  - Investigational Site Number 752002, Malmo
  - Investigational Site Number 752003, Skene
  - Investigational Site Number 752001, Stockholm
- Investigational Site Number 756001, Geneva, Switzerland
- Thailand (6):
  - Investigational Site Number 764004, Bangkok
  - Investigational Site Number 764001, Bangkok
  - Investigational Site Number 764002, Chiang Mai
  - Investigational Site Number 764003, Khon Kaen
  - Investigational Site Number 764006, Nakhonratchasima
  - Investigational Site Number 764005, Pathum Thani
- Investigational Site Number 784-001, Dubai, United Arab Emirates

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Home PD, Bolli GB, Mathieu C, Deerochanawong C, Landgraf W, Candelas C, Pilorget V, Dain MP, Riddle MC. Modulation of insulin dose titration using a hypoglycaemia-sensitive algorithm: insulin glargine versus neutral protamine Hagedorn insulin in insulin-naive people with type 2 diabetes. Diabetes Obes Metab. 2015 Jan;17(1):15-22. doi: 10.1111/dom.12329. Epub 2014 Jul 12. PMID 24957785